CLINICAL TRIAL: NCT06269432
Title: Precise Antiplatelet THerapy Guided by Platelet Aggregation Function in Ischemic STROKE
Brief Title: Precise Antiplatelet THerapy Guided by Platelet Aggregation Function in Ischemic STROKE（PATH-STROKE）
Acronym: PATH-STROKE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Jie Yang, Deputy Director of the Institute of Neurology, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023YFS0042
Record Dates: First submitted 2024-01-29; First posted 2024-02-21 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Ischemic Stroke; Antiplatelet Drug
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Precision Antiplatelet Therapy Trial Group (Experimental): Platelet function testing guides antiplatelet drug selection
  Interventions: Drug: Precision Antiplatelet Therapy Trial Group
- Traditional Antiplatelet Therapy Control Group (Active Comparator): Aspirin 100mg orally once a day
  Interventions: Drug: Traditional Antiplatelet Therapy Control Group

INTERVENTIONS:
Drug: Precision Antiplatelet Therapy Trial Group — Use SPCM method to detect platelet aggregation function in patients, adjust antiplatelet drugs based on the test results, and receive precise antiplatelet treatment for 12 months. Non resistant patients with aspirin will continue to receive aspirin 100mg qd; Patients with aspirin resistance were given clopidogrel 75mg qd; Clopidogrel resistant patients were given ticagrelor 90mg bid.
  Arms: Precision Antiplatelet Therapy Trial Group
Drug: Traditional Antiplatelet Therapy Control Group — No adjustment of antiplatelet medication is required, and routine treatment with aspirin 100mg qd is given for 12 months.
  Arms: Traditional Antiplatelet Therapy Control Group

SUMMARY:
1. Main objective: To explore the efficacy of precise antiplatelet therapy guided by platelet aggregation function in reducing the incidence of 30 day platelet hyperresponsiveness in patients with non-cardiogenic ischemic stroke.
2. Secondary objective: To explore the efficacy and safety of antiplatelet therapy in patients with non-cardiogenic ischemic stroke under the guidance of platelet aggregation function.

DETAILED DESCRIPTION:
Non cardiac cerebral infarction accounts for more than 50% of cerebral infarction cases, and the key to its onset is increased platelet aggregation function. Aspirin and clopidogrel are Class A recommended drugs for the prevention and treatment of non cardiac cerebral infarction. However, after regular use of aspirin and clopidogrel, more than 30% of stroke patients still experience high on treatment platelet reactivity (HOPR) due to aspirin resistance and clopidogrel resistance, leading to stroke recurrence. Antiplatelet therapy is the cornerstone of the prevention and treatment of non cardiogenic cerebral infarction. Therefore, clinical research on the prevention and treatment of HOPR with antiplatelet therapy for non cardiogenic cerebral infarction is of great significance, which can help partially solve the bottleneck of resistance to antiplatelet therapy in cerebral infarction.Platelet aggregation function testing can timely detect antiplatelet therapy HOPR, guide drug adjustment, and is expected to become a testing standard for the prevention and treatment of antiplatelet therapy resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18 to 80 years;
2. Diagnosed with non-cardiogenic ischemic stroke according to WHO criteria, confirmed by cranial CT or MRI to exclude hemorrhagic stroke.;
3. First stroke onset ≥ 1 month and ≤ 3 months;
4. mRS Score <=2 points;
5. Undergoing antiplatelet therapy with 100mg aspirin daily for at least 8 days;
6. Informed consent signed by the patient or their family member.

Exclusion Criteria:

1. History of recurrent stroke.
2. History of gastrointestinal bleeding, intracranial hemorrhage, or other bleeding disorders.
3. Contraindications or intolerance to antiplatelet therapy medications.
4. Severe cardiac, pulmonary, hepatic, or renal insufficiency, or presence of severe comorbid conditions (e.g., end-stage malignant tumors, severe single/multiple organ failure).
5. Poor compliance, inability to cooperate with study requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of HOPR at 30 ± 5 days post-enrollment. | 1-month
  The incidence of HOPR at 30 ± 5days post-enrollment.

SECONDARY OUTCOMES:
The occurrence of major ischemic events and major bleeding events. | 3-month
  Including cardiovascular and cerebrovascular death, myocardial infarction, stroke, urgent revascularization, in-stent thrombosis, and bleeding events classified as BARC grade 2 or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yang, doctor, Study Chair — Sichuan Provincial People's Hospital; YaPeng Lin, Study Chair — First Affiliated Hospital of Chengdu Medical College
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang W, Jiang B, Sun H, Ru X, Sun D, Wang L, Wang L, Jiang Y, Li Y, Wang Y, Chen Z, Wu S, Zhang Y, Wang D, Wang Y, Feigin VL; NESS-China Investigators. Prevalence, Incidence, and Mortality of Stroke in China: Results from a Nationwide Population-Based Survey of 480 687 Adults. Circulation. 2017 Feb 21;135(8):759-771. doi: 10.1161/CIRCULATIONAHA.116.025250. Epub 2017 Jan 4. PMID 28052979
- [Background] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Background] Liu L, Wang D, Wong KS, Wang Y. Stroke and stroke care in China: huge burden, significant workload, and a national priority. Stroke. 2011 Dec;42(12):3651-4. doi: 10.1161/STROKEAHA.111.635755. Epub 2011 Nov 3. PMID 22052510
- [Background] Mastenbroek TG, van Geffen JP, Heemskerk JW, Cosemans JM. Acute and persistent platelet and coagulant activities in atherothrombosis. J Thromb Haemost. 2015 Jun;13 Suppl 1:S272-80. doi: 10.1111/jth.12972. PMID 26149036
- [Background] Franchi F, Rollini F, Angiolillo DJ. Antithrombotic therapy for patients with STEMI undergoing primary PCI. Nat Rev Cardiol. 2017 Jun;14(6):361-379. doi: 10.1038/nrcardio.2017.18. Epub 2017 Feb 23. PMID 28230176
- [Background] Estevez B, Du X. New Concepts and Mechanisms of Platelet Activation Signaling. Physiology (Bethesda). 2017 Mar;32(2):162-177. doi: 10.1152/physiol.00020.2016. PMID 28228483
- [Background] Galli M, Benenati S, Capodanno D, Franchi F, Rollini F, D'Amario D, Porto I, Angiolillo DJ. Guided versus standard antiplatelet therapy in patients undergoing percutaneous coronary intervention: a systematic review and meta-analysis. Lancet. 2021 Apr 17;397(10283):1470-1483. doi: 10.1016/S0140-6736(21)00533-X. PMID 33865495
- [Background] Zheng YY, Wu TT, Yang Y, Hou XG, Gao Y, Chen Y, Yang YN, Li XM, Ma X, Ma YT, Xie X. Personalized antiplatelet therapy guided by a novel detection of platelet aggregation function in stable coronary artery disease patients undergoing percutaneous coronary intervention: a randomized controlled clinical trial. Eur Heart J Cardiovasc Pharmacother. 2020 Jul 1;6(4):211-221. doi: 10.1093/ehjcvp/pvz059. PMID 31603191
- [Background] Cayla G, Cuisset T, Silvain J, Leclercq F, Manzo-Silberman S, Saint-Etienne C, Delarche N, Bellemain-Appaix A, Range G, El Mahmoud R, Carrie D, Belle L, Souteyrand G, Aubry P, Sabouret P, du Fretay XH, Beygui F, Bonnet JL, Lattuca B, Pouillot C, Varenne O, Boueri Z, Van Belle E, Henry P, Motreff P, Elhadad S, Salem JE, Abtan J, Rousseau H, Collet JP, Vicaut E, Montalescot G; ANTARCTIC investigators. Platelet function monitoring to adjust antiplatelet therapy in elderly patients stented for an acute coronary syndrome (ANTARCTIC): an open-label, blinded-endpoint, randomised controlled superiority trial. Lancet. 2016 Oct 22;388(10055):2015-2022. doi: 10.1016/S0140-6736(16)31323-X. Epub 2016 Aug 28. PMID 27581531
- [Background] Zhu HC, Li Y, Guan SY, Li J, Wang XZ, Jing QM, Wang ZL, Han YL. Efficacy and safety of individually tailored antiplatelet therapy in patients with acute coronary syndrome after coronary stenting: a single center, randomized, feasibility study. J Geriatr Cardiol. 2015 Jan;12(1):23-9. doi: 10.11909/j.issn.1671-5411.2015.01.003. PMID 25678901
- [Background] Yi X, Lin J, Wang C, Huang R, Han Z, Li J. Platelet function-guided modification in antiplatelet therapy after acute ischemic stroke is associated with clinical outcomes in patients with aspirin nonresponse. Oncotarget. 2017 Nov 7;8(63):106258-106269. doi: 10.18632/oncotarget.22293. eCollection 2017 Dec 5. PMID 29290946